CLINICAL TRIAL: NCT04748536
Title: A Randomised, Double-blind, Placebo-controlled, Parallel Group Study in Healthy Volunteers to Assess the Safety, Tolerability and Pharmacokinetics of Multiple Ascending Doses of IRL201104 to Support a Future COVID-19 Patient Study
Brief Title: Safety and PK of Repeated Doses of IRL201104 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Revolo Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C1104-003
Record Dates: First submitted 2021-02-01; First posted 2021-02-10 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-02

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — IRL201104

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Dose A IRL201104 or placebo (Experimental): IRL201104 IV once daily for 5 days OR Placebo IV once daily for 5 days
  Interventions: Drug: IRL201104; Drug: Placebo
- Group 2: Dose B IRL201104 or placebo (Experimental): IRL201104 IV once daily for 7 days OR Placebo IV once daily for 7 days
  Interventions: Drug: IRL201104; Drug: Placebo

INTERVENTIONS:
Drug: IRL201104 — lyophilised powder for reconstitution for IV dosing
Drug: Placebo — Matching placebo for IRL201104

SUMMARY:
The purpose of this study is to assess the safety, tolerability and pharmacokinetics of repeat doses of IRL201104 given to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects age 18 to 65 years of age, and in good health as determined by medical history, physical examination, vital signs, electrocardiogram, and laboratory tests.
* Female subjects agree to use highly effective contraception or be of non-childbearing potential.
* Written informed consent must be obtained before any assessment is performed.
* Able to communicate well with the Investigator/designee.

Exclusion Criteria:

* Any known reaction to study drug or components
* concurrent or recent infection or clinically significant conditions that may place subject at risk or interference with absorption, distribution or excretion of drugs
* No QTcF interval ≥450 milliseconds, no QRS complex ≥120 milliseconds, at Screening
* Positive test results for hepatitis B surface antigen (HBsAg), hepatitis C virus antibodies (HCVAb) or human immunodeficiency virus (HIV) 1 and/or -2 antibodies at Screening.
* Excessive use of caffeine-containing beverages
* Urinary cotinine level indicative of smoking or history or regular use of tobacco- or nicotine containing products within 6 months before screening.
* Presence or history of drug of alcohol abuse.
* Positive screen for drugs-of-abuse or cotinine.
* Blood donation in excess of 500mL within 3 months.
* Participation in another clinical study with licensed or unlicensed study drug within 3 months of first IMP administration.
* Exposure to more than 4 new chemical entities within 12 months before the first IMP administration.
* Use of live vaccine 28 days before dosing with study drug until telephone follow-up and use of killed vaccine (including COVID-19 vaccine) 14 days before dosing with study drug until telephone follow-up.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2021-04-05 (Actual); Study Completion 2021-04-05 (Actual)

PRIMARY OUTCOMES:
Number of subjects with TEAEs and number of events will be summarised by treatment | 33 (group 1) or 35 (group 2) days
  Adverse Events after treatment administration will be collected at baseline and repeated until study completion
Number of subjects with potentially clinically important (PCI) abnormal haematology variables will be summarised by treatment | 19 (group 1) or 21 (group 2) days
  Haemoglobin, haematocrit, MCV, MCH, MCHC, RBC, WBC and differentials will be collected at baseline and after dose administration and repeated until Day 19 or 21
Number of subjects with PCI abnormal clinical chemistry variables will be summarised by treatment | 19 (group 1) or 21 (group 2) days
  Creatinine, glucose, triglycerides, urea, uric acid, bilirubin, cholesterol, sodium, potassium, alkaline phosphatase, AST, ALT and GGT will be collected at baseline and after dose administration and repeated until Day 19 or 21
Number of subjects with PCI and/or abnormal electrocardiogram variables will be summarised by treatment | 19 (group 1) or 21 (group 2) days
  RR, PR, QRS, QT-interval, QTcF and heart rate will be collected at baseline and after dose administration and repeated until Day 19 or 21.
Number of subjects with PCI abnormal vital sign variables will be summarised by treatment | 19 (group 1) or 21 (group 2) days
  Blood pressure, pulse rate, oral body temperature and respiration rate will be collected at baseline and after single and multiple dose administration and repeated until Day 19 or 21

SECONDARY OUTCOMES:
Pharmacokinetics of IRL201104: Trough blood concentration (Ctrough) | 5 (group 1) or 7 (group 2) days
  Ctrough will be measured after multiple dosing
PK of IRL201104: Maximum (peak) blood concentration (Cmax) | 5 (group 1) or 7 (group 2) days
  Cmax will be calculated after multiple dosing
PK of IRL201104: Terminal half life (t1/2) | 5 (group 1) or 7 (group 2) days
  t1/2 will be calculated after multiple dosing
PK of IRL201104: Area under the curve from time zero to last quantifiable concentration of IRL201104 (AUCt) | 5 (group 1) or 7 (group 2) days
  AUCt will be calculated after multiple dosing
PK of IRL201104: Apparent total body clearance from blood (CLss) | 5 (group 1) or 7 (group 2) days
  CLss will be calculated after multiple dosing
PK of IRL201104: steady state volume of distribution (Vz) | 5 (group 1) or 7 (group 2) days
  Vz will be calculated after multiple dosing

CONTACTS AND LOCATIONS:
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom